CLINICAL TRIAL: NCT01602328
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Study of AC607 for the Treatment of Acute Kidney Injury in Cardiac Surgery Subjects
Brief Title: A Study to Evaluate the Safety and Efficacy of AC607 for the Treatment of Kidney Injury in Cardiac Surgery Subjects
Acronym: ACT-AKI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AlloCure Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC 6071103
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Acute renal failure; Human mesenchymal stem cells; Allogeneic stem cells
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC607 (Active Comparator): Treatment with AC607
  Interventions: Biological: AC607
- Placebo (Placebo Comparator): Treatment with Placebo
  Interventions: Biological: Vehicle Only

INTERVENTIONS:
Biological: AC607 — AC607 will be a single administration at a target dose of 2 x 10E6 hMSC/kg body weight
  Other Names: allogeneic bone marrow-derived human mesenchymal; stem cells
  Arms: AC607
Biological: Vehicle Only — The dose will be calculated and recorded in the same way as for AC607.
  Arms: Placebo

SUMMARY:
Subjects entering the study will have undergone cardiac surgery. Those who experience kidney injury within 48 hours of their surgery will be enrolled into the study. Once enrolled, subjects will receive a single administration of AC607 or placebo. Kidney recovery will be evaluated over the subsequent 30 days and death or the need for dialysis will be evaluated within 90 days of dosing. After 90 days (evaluation period), subjects will enter a 3-year extension phase of the study to monitor safety and long-term outcomes (follow-up period).

DETAILED DESCRIPTION:
The study will enroll post-cardiac surgery subjects (CABG and/or valve) with laboratory evidence of AKI within 48 hrs of removal from cardiopulmonary bypass. Subjects will be randomly assigned (1:1 ratio) to treatment with a single administration of AC607 or placebo (approximately 100 subjects per group).

Safety and efficacy assessments will be performed daily during the post-operative hospital stay from the day randomized into the study until discharge, at 30 days, and at 90 days after study drug administration (evaluation phase). Safety and long-term clinical outcomes will be assessed at 6, 12, 24 and 36 months (long-term follow-up phase).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Had cardiovascular surgery utilizing cardiopulmonary bypass
* Have a pre-operative (baseline) serum creatinine value collected within 30 days of surgery (if multiple laboratory results are available within this time window, the most recent serum creatinine value prior to surgery will be used to establish the baseline)
* Willing and able to comply with visit schedule and study procedures including post-hospitalization discharge follow-up
* Ability to give informed consent or have a legally acceptable representative do so for them
* Have AKI defined as ≥ 0.5 mg/dL rise in serum creatinine from baseline within 48 hours of removal from cardiopulmonary bypass

Exclusion Criteria:

* Active cancer and/or receiving active treatment for cancer, with the exception of squamous cell or basal cell carcinoma of the skin
* Had surgery for thoraco-abdominal aortic aneurysm (TAAA)
* Currently participating in another interventional drug or device clinical study
* Prisoner or other detainee
* Has a current medical condition that would preclude or compromise femoral artery catheter placement
* Has an intra-aortic balloon pump (IABP) in place within 2 hours of catheter placement
* Has a ventricular assist device (VAD) or extracorporeal membrane oxygenation (ECMO) in place at the time of the study catheter placement
* Prior history of solid organ or bone marrow transplant
* Stage 5 CKD or currently on dialysis
* Are expected to receive dialysis within 24 hours of enrollment or dosing
* Had a complication during surgery or post-operatively that, in the opinion of the principal investigator (PI), significantly increases the risk of complications to the subject and therefore precludes dosing the subject
* Are pregnant or lactating. A woman with child-bearing potential may be tested for pregnancy at the discretion of the PI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time to Kidney Recovery defined as a post-operative serum creatinine return to pre-operative baseline values. | Within 30 days of dosing.
  The first occurrence of a post-dosing serum creatinine level that is equal to or less than the subject's pre-operative baseline level.

SECONDARY OUTCOMES:
All-Cause Mortality or Dialysis (composite endpoint). | Subjects who died or received dialysis within 30 and 90 days after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Viken Paragamian, Study Director
Locations (31):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Stanford Hospital and Clinics, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - UTHealth, The University of Texas Health Science Center at Houston, Houston, Texas
  - Fletcher Allen Health Care - Renal Services, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Manitoba - St. Boniface Hospital, Winnipeg, Manitoba
  - CDHA Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster - Hamilton General Hospital / TAARI, Hamilton, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Zhao L, Hu C, Zhang P, Jiang H, Chen J. Preconditioning strategies for improving the survival rate and paracrine ability of mesenchymal stem cells in acute kidney injury. J Cell Mol Med. 2019 Feb;23(2):720-730. doi: 10.1111/jcmm.14035. Epub 2018 Nov 28. PMID 30484934